CLINICAL TRIAL: NCT02878850
Title: Randomized Trial of Early Hemodynamic Management of Patients Following Acute Spinal Cord Injury
Acronym: TEMPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miriam Treggiari, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEMPLE - 001; CDMRP-SC150250 (Other Grant/Funding Number: United States Department of Defense, CDMRP)
Record Dates: First submitted 2016-08-03; First posted 2016-08-25 (Estimated); Results first posted 2025-11-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Blood Pressure (Experimental): Subjects will have their blood pressure kept in a higher range.
  Interventions: Other: Augmented Blood Pressure
- Conventional Blood Pressure (No Intervention): Subjects will have their blood pressure kept in a normal range.

INTERVENTIONS:
Other: Augmented Blood Pressure — Subjects will have their blood pressure kept in a higher range.
  Arms: Augmented Blood Pressure

SUMMARY:
The purpose of this study is to learn more about how participants heal from acute spinal cord injury.

DETAILED DESCRIPTION:
In this study, the investigators will learn about the effect of targeted blood pressure management (TPM) on participants healing from acute spinal cord injury.

The investigators want to learn:

The effect of two types of TPM on long term motor and sensory outcomes. The effect of two types of TPM on long-term pain and functional independence outcomes.

How safe TPM is for participants.

ELIGIBILITY:
Inclusion Criteria:

1. Acute traumatic spinal cord injury (SCI) involving neurological levels as defined by the ASIA neurological examination between C0 and T8 (tetraplegia) and resulting in new onset neurological deficits consistent with an ASIA motor assessment of level A, B or C.
2. Subject is 18 years of age or older.

Exclusion Criteria:

1. Penetrating SCI injury.
2. Isolated cauda equina syndrome or injury at bony level Th9 or below.
3. Pre-existing motor deficit secondary to chronic myelopathy.
4. History of demyelinating disease or central nervous system autoimmune disorder.
5. History within the past six months and/or physical findings on admission of decompensated congestive heart failure (NYHA functional class III or IV, or objective class C or D).
6. Acute, evolving or recent (30 days) myocardial infarction.
7. Chronic renal failure requiring dialysis.
8. Suspected or confirmed pregnancy.
9. Severe terminal disease with life expectancy less than 6 months.
10. Severe traumatic brain injury at presentation (GCS ≤8) with confirmation of injury on brain imaging.
11. A condition that would preclude the performance of an accurate neurological exam due to a prior diagnosis of Alzheimer's disease, stroke, degenerative condition, cerebral tumor, or mental retardation.
12. Non-English or Non-Spanish Speaking.
13. Refusal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, PhD, MPH, Principal Investigator — Oregon Health and Science University
Locations (11):
- United States (11):
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Atrium Health F.H. Sammy Ross Trauma Center, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sajdeya R, Yanez ND, Kampp M, Goodman MD, Zonies D, Togioka B, Nunn A, Winfield RD, Martin ND, Kohli A, Huynh TT, Okonkwo DO, Poblete RA, Gilmore EJ, Chesnut RM, Bunnell AE, Ohnuma T, Hashemaghaie M, Treggiari MM. Early Blood Pressure Targets in Acute Spinal Cord Injury: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2525364. doi: 10.1001/jamanetworkopen.2025.25364. PMID 40965887
- [Derived] Weinberg JA, Farber SH, Kalamchi LD, Brigeman ST, Bohl MA, Varda BM, Sioda NA, Radosevich JJ, Chapple KM, Snyder LA. Mean arterial pressure maintenance following spinal cord injury: Does meeting the target matter? J Trauma Acute Care Surg. 2021 Jan 1;90(1):97-106. doi: 10.1097/TA.0000000000002953. PMID 33003016

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Started | 46 | 46
Completed | 30 | 35
Not Completed | 16 | 11

BASELINE CHARACTERISTICS:
Population: 1 participant in the ABP and 1 participant in the CBP group were excluded due to inadequate consent documentation
Groups:
- Total: Total of all reporting groups
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (17.8) | 54.0 (17.9) | 53.8 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 38 | 38 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 7 | 5 | 12
Baseline American Spinal Injury Association (ASIA) Score [Mean (Standard Deviation); unit: Score] — The ASIA Score has a motor and a sensory component. The maximum Upper Extremities Motor Score (UEMS) is 50, the maximum Lower Extremities Motor Score (LEMS) is 50, the maximum Total Sensory Score (sum of pin prick [max 112] and light touch [max 112]) is 224. The minimum score is 0. Higher scores indicate better neurological outcome. Population: A complete neurological exam could not be obtained in 3 patients
  Score
    Upper Extremities Motor Score: number analyzed (Participants) | 46 | 43 | 89
    Upper Extremities Motor Score | 17.1 (13.4) | 23.0 (17.8) | 19.2 (15.9)
    Lower Extremities Motor Score: number analyzed (Participants) | 46 | 43 | 89
    Lower Extremities Motor Score | 6.9 (13.6) | 6.1 (12.2) | 6.5 (12.8)
    Total Sensory Score: number analyzed (Participants) | 46 | 43 | 89
    Total Sensory Score | 87.8 (54.4) | 77.3 (44.2) | 82.7 (49.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in American Spinal Injury (ASIA) Upper Extremities Motor Score
Description: Change from baseline in ASIA Upper Extremities Motor Score (UEMS), comparing patients maintained at a MAP target between 65 and 70 mm Hg, and patients maintained at a MAP target between 85 and 90 mm Hg for a duration of seven days or until ICU discharge. The UEMS score ranges from 0 to 50, with 50 indicating no deficits.
Time Frame: 6 months after spinal cord injury
Population: ABP: 46 patients allocated to intervention, 8 died, 3 unable to complete physical exam, 16 lost to follow up CBP: 46 patients allocated to intervention, 7 died, 9 unable to complete physical exam, 11 lost to follow up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 19 | 19
Scores on a scale | 15.58 (16.23) | 12.63 (13.42)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = 2.95, 95% CI 2-sided [-6.85 to 12.75]

2. Secondary Outcome: Spinal Cord Independence Measure III Score
Description: Spinal Cord Independence Measure III (SCIM III). The total SCIM III Score ranges from 0 to 100 points, with 0 indicating complete dependence and 100 indicating complete independence.
Time Frame: 6 months after spinal cord injury
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 22 | 26
Scores on a scale | 27.48 (19.43) | 28.11 (20.82)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.92, ANCOVA; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-12.48 to 11.21]

3. Secondary Outcome: Pain Scores on the International Spinal Cord Injury Basic Pain Data Set
Description: Pain Interference with daily activity on the International Spinal Cord Injury Basic Pain Data Set. Pain Interference Score ranges from 0 to 10, with higher scores indicating higher pain levels.
Time Frame: 6 months after spinal cord injury
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 22 | 26
Scores on a scale | 5.21 (3.17) | 4.86 (3.66)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.75, ANCOVA; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-1.83 to 2.53]

4. Secondary Outcome: International Spinal Cord Injury Quality of Life (ISCIQoL) Basic Data Set
Description: The ISCIQoL Basic Data Set is a 3-item self-report tool of quality of life across three domains: 1. Satisfaction with life as a whole; 2. Satisfaction with physical health; 3. Satisfaction with psychological health. Each domain scores from 0 to 10, and the total score range (sum of the 3 domains) ranges from 0 to 30. Higher scores indicate better perceived quality of life.
Time Frame: 6 months after spinal cord injury
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 22 | 26
Scores on a scale | 19.94 (6.43) | 18.00 (7.31)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.40, ANCOVA; Mean Difference (Final Values) = 1.94, 95% CI 2-sided [-2.64 to 6.53]

5. Other Pre Specified Outcome: Incidence of Respiratory Complications
Description: Incidence of respiratory complications
Time Frame: 7 days after randomization or ICU discharge, whichever came first, assessed up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 45 | 45
Participants | 36 | 18
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p < 0.001, Chi-squared; Risk Ratio (RR) = 2.00, 95% CI [1.36 to 2.94]

6. Other Pre Specified Outcome: Cardiovascular Function
Description: Hypotension, hypertension, autonomic dysreflexia, edema, pulmonary embolism, deep venous thrombosis, other cardiovascular condition.
Time Frame: 6 months after spinal cord injury
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 19 | 24
Participants | 6 | 7
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.87, Chi-squared; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.44 to 3.65]

7. Other Pre Specified Outcome: Sequential Multiple Organ Assessment (SOFA) Score
Description: Modified Sequential Multiple Organ Assessment (SOFA) score on Day 7 after randomization. The modified SOFA score does not include the points contributed by the Cardiovascular system. The modified SOFA score ranges from 0 to 20, with higher scores indicating greater organ dysfunction and higher mortality risk.
Time Frame: 7 days after randomization
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 43 | 40
Scores on a scale | 1.40 (1.84) | 0.78 (1.33)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.08, ANCOVA; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.08 to 1.32]

8. Primary Outcome: Change From Baseline in American Spinal Injury (ASIA) Lower Extremities Motor Score
Description: Change from baseline in ASIA Lower Extremities Motor Score (LEMS), comparing patients maintained at a MAP target between 65 and 70 mm Hg, and patients maintained at a MAP target between 85 and 90 mm Hg for a duration of seven days or until ICU discharge. The LEMS score ranges from 0 to 50, with 50 indicating no deficits.
Time Frame: 6 months after spinal cord injury
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 19 | 19
Scores on a scale | 10.79 (16.66) | 16.16 (18.16)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.35, t-test, 2 sided; Mean Difference (Final Values) = -5.73, 95% CI 2-sided [-16.84 to 6.10]

9. Primary Outcome: Change From Baseline in American Spinal Injury Association (ASIA) Sensory Score
Description: Change from baseline in ASIA Sensory Score, comparing patients maintained at a MAP target between 65 and 70 mm Hg, and patients maintained at a MAP target between 85 and 90 mm Hg for a duration of seven days or until ICU discharge. The total Sensory Score adds light touch points (max 112) and pin prick points (max 112). The total score ranges from 0 to 224, with higher scores indicating better neurological outcomes.
Time Frame: 6 months after spinal cord injury
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
Number analyzed (Participants) | 19 | 19
Scores on a scale | 6.26 (41.32) | 41.63 (58.97)
Statistical Analysis 1: Comparison: Augmented Blood Pressure vs Conventional Blood Pressure; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = -35.37, 95% CI 2-sided [-68.87 to -1.87]

ADVERSE EVENTS:
Time Frame: From enrollment up to 6 months
Arm/Group | Augmented Blood Pressure | Conventional Blood Pressure
All-Cause Mortality (participants affected / at risk) | 8/46 | 7/46
Serious Adverse Events (participants affected / at risk) | 12/46 | 13/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Augmented Blood Pressure (N=46) | Conventional Blood Pressure (N=46)
Cardiac Arrest (Cardiac disorders) | 3 (3) | 5 (5)
Respiratory Complications (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Sepsis/Infection (Infections and infestations) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT02878850/Prot_SAP_000.pdf